CLINICAL TRIAL: NCT04965688
Title: Systems Biology Guided Therapy for Breast Cancer Positive for Oestrogen Receptor After Aromatase Inhibitor and CDK Inhibition
Brief Title: Biology Guided Therapy for Breast Cancer for ER Positive
Acronym: SPOCK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment to meet the primary and secondary study goals
Sponsor: Inova Health Care Services (Other)
Collaborators: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U21-02-4401
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Cancer Treatment Based on Biopsy Results (Other)
  Interventions: Drug: Biopsy-Guided Therapy Selection

INTERVENTIONS:
Drug: Biopsy-Guided Therapy Selection — All enrolled participants will undergo a tumor biopsy, which will be analyzed for genomic and transcriptomic alterations using FoundationOne (DNA) and Fulgent (RNA). Based on the genomic findings, participants will receive one of the following therapy standard-of-care treatment options:
  PI3K inhibitor + anti-estrogen therapy ( alpelisib + fulvestrant)
  MTOR inhibitor + anti-estrogen therapy (everolimus + exemestane)
  Anti-estrogen therapy alone (fulvestrant monotherapy)
  Cytotoxic chemotherapy (capecitabine)

SUMMARY:
There are several approved and guideline-recommended treatments for metastatic, estrogen receptor-positive breast cancer that has progressed on an aromatase inhibitor and a CDK4/6 inhibitor. Right now, doctors do not have a good way of choosing between these treatments. Scientists we work with have come up with ways to use the biology of the tumor to try to predict which treatment is best. This study is being done to test if those predictions are right and to learn more about these tumors to design better treatments in the future.

DETAILED DESCRIPTION:
This is an open-label phase II study of systems biology guided therapy for breast cancer patients positive for Oestrogen receptor after Aromatase inhibitor and CDK inhibition.

Based on the SOLAR-1 trial, 25% of tumors would have PIK3CA mutation, so 25% of people would be treated with fulvestrant plus alpelisib with a median PFS in that group of 11 months and 75% of people would be treated with fulvestrant with a median PFS in that group of 6 months.(3) The weighted average of these medians is 7.25 months, but since the actual distributions of the progression free survivals are not available, we will use a conservative estimate of the expected median PFS of the historical control group (fulvestrant +/- alpelisib as second line unguided therapy) of 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of breast cancer
* Metastatic or incurable
* Prior treatment with an anastrozole or letrozole and a CDK4/6 inhibitor
* Progression while on or within 6 months of stopping the CDK4/6 inhibitor
* At least one lesion amenable to percutaneous biopsy that is not a purely sclerotic bone lesion
* ECOG 0-2
* Age 18 or greater
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior treatment within 2 years with fulvestrant, alpelisib, everolimus, or capecitabine
* Comorbid disease other than breast cancer with a life expectancy of less than 2 years
* Cancer other than breast cancer that is expected to need treatment within 2 years
* Platelets < 100,000/microliter
* INR > 1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cohen, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aromatase Inhibitor and CDK Inhibition: Drug determined by treating oncologist based on recommendation from systems biology analysis.: All patients will have a biopsy at the beginning of the trial. The biopsy will be sent for DNA sequencing through FoundationOne(clinical test) and RNA profiling at Fulgent(research test) for determination of activation of various oncogenic pathways and phenotypes. The results will be analyzed and a treatment recommendation will be made to the treating physician based on an algorithm.
Period: Overall Study
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Baseline to 36 Months
Population: Two patients enrolled on the study and then withdrew early prior to treatment, therefore no data were collected before study termination.
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Number analyzed (Participants) | 0

2. Secondary Outcome: Turn Around Time for Systems Biology Analysis
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Baseline to 36 Months
Population: as for outcome 1
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate to Systems Biology Guided Therapy
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Baseline to 36 Months
Population: as for outcome 1
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival Base on Concordance With Recommended Treatment
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Baseline to 36 Months
Population: as for outcome 1
Arm/Group | Aromatase Inhibitor and CDK Inhibition
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to 36 months.
Arm/Group | Aromatase Inhibitor and CDK Inhibition
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04965688/Prot_SAP_ICF_001.pdf